CLINICAL TRIAL: NCT06070805
Title: The Impact and Mechanism of Depression on Cardio-cerebral Vascular Events and Arteriovenous Fistula Dysfunction in Hemodialysis Patients: A Single Center and Real-world Study
Brief Title: Impact and Mechanism of Depression on Cardio-cerebral Vascular Events and Arteriovenous Fistula Dysfunction in MHD Patients
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Yunfeng Xia, Clinical Professor, First Affiliated Hospital of Chongqing Medical University
Other Study IDs: 1st ChongqingMU
Record Dates: First submitted 2023-10-02; First posted 2023-10-06 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Cardio-cerebral Vascular Events; Arteriovenous Fistula Dysfunction
Keywords: maintenance hemodialysis patients; depression; cardio-cerebral vascular events; arteriovenous fistula dysfunction; platelet
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-depression group: The Hamilton Rating Scale for Depression (HAMD) will be applied to assess the depressive status of all enrolled patients. This scale consists of 24 survey items, each with a score of 0-4. Patients will be assigned to the nondepression group if their HAMD score was <8.
  Interventions: Other: depression
- Depression group: Patients will be assigned to the depression group if their score was ≥8.
  Interventions: Other: depression

INTERVENTIONS:
Other: depression — The score of Hamilton Rating Scale for Depression (HAMD) is ≥8

SUMMARY:
Depression is a common psychiatric disorder in patients on maintenance hemodialysis (MHD). It may contribute to poor prognosis in a number of ways, including its effect on platelet function. We aimed to investigate the impact and underlying mechanisms of depression on the occurrence of cardio-cerebral vascular events (CCVE) and dysfunction of arteriovenous fistula (DAVF) in MHD patients.

In this study, MHD patients were recruited and divided into depression and non-depression groups using the Hamilton Depression Scale (HAMD) in this prospective cohort study. Their clinical and laboratory indicators were collected and the occurrence of CCVE and DAVF were recorded through clinical follow-up, and analyzed, and the differences and possible influencing factors of CCVE and DAVF occurrence were assessed between the two groups of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients had undergone dialysis treatment for more than 3 months, and their medical status was stable at the time of enrollment, with an expected survival period of more than 1 year

Exclusion Criteria:

* (1) with communication disorders or mental illness other than depression; (2) a combination of cirrhosis, lymphoma, thrombocytopenic purpura, or other diseases that significantly affect platelet function; (3) complicated with malignant tumors, tuberculosis, severe heart failure, and unstable medical conditions; (4) inability or unwillingness to cooperate with researchers.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing maintenance hemodialysis were recruited from the First Affiliated Hospital of Chongqing Medical University in China.
Sampling Method: Non-Probability Sample
Enrollment: 286 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-04-08 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
cardio-cerebral vascular events (CCVE) | 1 year
  CCVEs were defined as the first occurrence of angina pectoris, myocardial infarction, episodes of heart failure requiring clinical intervention, arrhythmic episodes with clinically significant symptoms, transient ischemic attack, cerebral infarction, and cerebral hemorrhage during the observational period.
dysfunction of arteriovenous fistula (DAVF) | 1 year
  DAVF was diagnosed if a patient presented with any one or more of the following conditions that render his or her AVF unsatisfactory for effective hemodialysis: (1) loss of AVF murmur on clinical auscultation; (2) notable weakening or disappearance of pulsation in AVF; (3) echography showing interruption of blood flow, thrombosis within the internal fistula, or stenosis of the venous outflow tract at or near the anastomotic site; or (4) maximum blood flow <200 mL/min in AVF during dialysis.

CONTACTS AND LOCATIONS:
Overall Officials: Yunfeng Xia, Dr, Study Director — First Affiliated Hospital of Chongqing Medical University
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided